CLINICAL TRIAL: NCT00391859
Title: Pharmacist-initiated Intervention Trial in OsteoArthritis (PhIT-OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Arthritis Network (Network); Michael Smith Foundation for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H06-70373; H06-70373
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
Keywords: Pharmacist-initiated Intervention Trial in OsteoArthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health service provision (Experimental): Health service provision within the first few months of diagnosis which includes physical examination, radiographs, education, exercise, weight loss, assistive devices and pharmacologic therapy.
  Interventions: Procedure: Pharmacist-Initiated Intervention in OsteoArthritis (PhIT-OA)

INTERVENTIONS:
Procedure: Pharmacist-Initiated Intervention in OsteoArthritis (PhIT-OA) — See Detailed Description.

SUMMARY:
Osteoarthritis (OA) is a major public health concern. Currently, there are at least 3 million Canadians afflicted with this condition with a 50% increase predicted by 2020. It is estimated that 85% of Canadians are afflicted with OA by age 70. As such, using the current health care structure, it is doubtful that the health system can keep pace with this increasing demand. Alternative health care delivery strategies must be investigated.

The purpose of this study is to assess if a pharmacist-initiated intervention for individuals with knee pain with a high likelihood of knee OA will lead to an improvement in the quality of care for these individuals.

We are hopeful that results of this study will show better management of knee osteoarthritis by a pharmacist-initiated intervention (which means that it is the pharmacist who will start the process for an intervention that includes exercise and an educational program when compared to no intervention. If this is the case, by implementing the proposed intervention program, subjects could be diagnosed earlier, the burden of illness on individuals could be diminished through an appropriate intervention program, and economic savings could be embraced.

Hypothesis: Community pharmacists can identify patients with likely knee OA and initiate a multidisciplinary intervention that will improve quality of care and outcomes.

DETAILED DESCRIPTION:
This will be a pilot study of a multidisciplinary intervention for individuals with knee pain with a high likelihood of knee OA that could be a model for other chronic diseases. The intervention will be multidisciplinary such that it will be initiated by community pharmacists with referral to a comprehensive OA treatment program at the provincial arthritis center involving physiotherapists. In addition, formal communication will be initiated with their family doctor. Those in the usual care group will receive an educational OA pamphlet. The primary objective of this pilot project is to determine the proportion of patients who meet the Arthritis Foundation's Quality Indicator Set for osteoarthritis in the treatment arm compared to those in the usual care arm. Specifically, this indicator set focuses on health service provision within the first few months of diagnosis which includes physical examination, radiographs, education, exercise, weight loss, assistive devices and pharmacologic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >50 years
2. ≥ 4 weeks of pain, aching or discomfort in or around the knee
3. Overweight or obese defined as BMI defined as ≥ 27 kg/m2
4. Not actively participating in a formal exercise program within the past 6 months
5. Self-reported difficulty in at least one of the following activities attributed to knee pain: lifting and carrying groceries, walking one quarter of a mile, getting in and out of a chair, or going up and down stairs.
6. Meet eligibility using the criteria on the pharmacist screening form (see attachment) - This form was adapted from the PhIND-OA study and amended to include points #3 to 6 above.

Exclusion Criteria:

1. Significant co-morbid disease that would pose a safety threat or impair ability to participate in an exercise program
2. Inability or unwillingness to modify dietary or exercise behaviours.
3. Knee X-Ray within the last 2 years
4. Inability to speak and write English
5. Knee pain due only to referred pain from osteoarthritis of the hip

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the difference in proportion of patients who receive ≥ 5 of the Arthritis Foundation's quality indicators during the six months of the study. | 6 months
(Baseline, months 2 and 6 ) | Months 2 and 6

SECONDARY OUTCOMES:
There are four secondary outcome measures that will be compared between intervention and usual care subjects at baseline, months 2 and 6: | Months 2 and 6
The difference in change of physical functioning (using the mean score from 17 questions from the WOMAC that are directed towards this construct) between intervention and usual care. This outcome has been used in recent, well-designed trials of OA.
The difference in knee pain (as assessed by five questions on the WOMAC);
The difference in Health Utilities Index Mark 3 (HUI3); and
The direct medical resource utilization using a questionnaire validated for use in musculoskeletal diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Marra, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Mary Pack Arthritis Center, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Marra CA, Cibere J, Grubisic M, Grindrod KA, Gastonguay L, Thomas JM, Embley P, Colley L, Tsuyuki RT, Khan KM, Esdaile JM. Pharmacist-initiated intervention trial in osteoarthritis: a multidisciplinary intervention for knee osteoarthritis. Arthritis Care Res (Hoboken). 2012 Dec;64(12):1837-45. doi: 10.1002/acr.21763. PMID 22930542